CLINICAL TRIAL: NCT04916626
Title: The OPUS YOUNG Study. The Efficacy of Early Intervention Service Versus Treatment as Usual for Adolescents Aged 12 - 17 With First-episode Psychosis, a Pragmatic Randomized Clinical Trial
Brief Title: The OPUS YOUNG Trial. Early Intervention Versus Treatment as Usual for Adolescents With First-episode Psychosis
Acronym: OPUS-YOUNG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Anne Katrine Pagsberg, Professor, PhD, senior consultant (child and adolescent psychiatry) and senior researcher., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPUS YOUNG
Record Dates: First submitted 2021-05-06; First posted 2021-06-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Schizotypal Disorder; Delusional Disorder; Acute and Transient Psychotic Disorder, Unspecified; Schizoaffective Disorder; Non-Organic Psychosis; Depression Severe; Substance Induced Psychoses
Keywords: Specialized early intervention; Early onset psychosis; Children and adolescents; Recovery and resilience; Cost-effectiveness; Cross-sectional
MeSH Terms: conditions — Schizophrenia; Schizotypal Personality Disorder; Schizophrenia, Paranoid; Psychotic Disorders; Mental Disorders; Psychoses, Substance-Induced | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The randomized clinical trial is a parallel, two-arm, superiority trial comparing OPUS YOUNG with TAU for children and adolescents aged 12 - 17 years with a first episode psychosis
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors are masked. The statistical evaluation of the effects of OY versus TAU will be carried out by researchers who will be masked for the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPUS YOUNG (Experimental): OPUS YOUNG is a two years out-patients specialized early intervention services for children and adolescents with a first episode psychosis. OPUS YOUNG is characterized by a multidisciplinary team, assertive outreach, tailored cognitive behavioral case management, and low caseload and insensitive psychoeducational family involvement
  Interventions: Behavioral: OPUS YOUNG
- Treatment as Usual, TAU (Active Comparator): Treatment as Usual will be carried out by outpatient clinic in Child and Adolescent Mental Health Services (CAMHS). Patients will be offered treatment following national Danish guidelines and local guidelines, provided by a multidisciplinary team, case-management (no defined upper-case load), family support. In general, office visits take place in outpatient clinics.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: OPUS YOUNG — OPUS YOUNG is a two year out-patient specialized early intervention service for children and adolescents with a first episode psychosis. The OPUS YOUNG treatment consists of the following elements: modified assertive community treatment, low patients to case manager ratio, cognitive-behavioural case management (CBCM), psycho-educational family treatment including multiple family groups(MFG) and psychoeducational siblings groups, Social Cognition and Interaction Training (SCIT), possible individual Cognitive Behavioural Therapy (CBT) in addition to CBCM, and manual based psychopharmacologic treatment. Additional, special transition support, individual school/employment support, and prevention and treatment of substance abuse.
  Arms: OPUS YOUNG
Behavioral: Treatment as Usual — The patients allocated to TAU will be offered non-manualized treatment following national Danish guidelines and local guidelines. Treatment is provided by a multidisciplinary team and consists of case-management (no defined upper case load), family support and psychoeducation, in addition to psychopharmacological treatment. In some cases, social skills training and CBT may be offered. In general, office visits take place in outpatient clinics.
  Arms: Treatment as Usual, TAU

SUMMARY:
The OPUS YOUNG (OY) study investigates the efficacy of early intervention service versus treatment as usual (TAU) for adolescents aged 12-17 years with a first-episode psychosis.

In Denmark, the yearly incidence of schizophrenia in youth below the age of 18 years has increased from 137 in 2000 to 477 in 2016. Outcomes in people with schizophrenia spectrum disorders are suboptimal with low quality of life, low rates of recovery, substance misuse, higher rates of suicide, violence and legal problems, low educational and vocational attainment, and a significantly reduced life-expectancy of 15-20 year. Schizophrenia imply a large burden of disease with severe impact on patients, their families, the service system and a large economic societal burden.

The investigators will include 290 participants age 12-17 years with an early onset psychosis within the following diagnostic classes: schizophrenia spectrum, psychotic depression or drug-induced psychosis. The design is an independent, investigator initiated, pragmatic, randomized clinical trial, with blinded outcome assessment. Participants are randomized 1:1 to OY or TAU. Participants in OY are offered 2 years of specialized intervention (OY) regardless of age, while participants in TAU are switched to adult psychiatry at the age of 18 years. OY builds on the Danish evidenced based intervention for young adults, OPUS, adjusted to meet the specific needs of adolescents: intensified support for caretakers and relatives including siblings; social cognition and interaction treatment; and individual cognitive behavioral case management. OY addresses the specific challenges of psychopharmacologic treatment in youth; supported transition to adult care after OY; school or educational support; and prevention and treatment of substance misuse. The primary endpoint is improved functioning in daily and social life after 24 months. Secondary outcome measures are psychopathology, quality of life, family stress, and retention in treatment and school/employment, and healthcare consumption. The clinical and societal perspective of a large scale implementation is improved prevention of the negative consequences of early-onset psychosis and a reduced burden of severe mental illness.

DETAILED DESCRIPTION:
The overarching purpose of the OPUS YOUNG trial is to improve the treatment and outcome of first-episode psychosis (FEP) in children and adolescents. We will address this ambition by testing the hypothesis, that Early Intervention Services (EIS) is superior compared to standard care in the treatment of children and adolescents below age 18 years with first-episode psychosis. The hypothesis is based on extrapolation of research showing that EIS is superior to standard care in the treatment of adults with first-episode psychosis with regards to symptom reduction, function improvement, adherence to treatment, lower hospitalization risk, improved recovery, and higher cost-effectiveness. However, no trials have investigated EIS in samples of patients below age 18 years. We will compare the efficacy and cost-effectiveness of EIS to treatment as usual (TAU) in adolescents aged 12-17 years (both inclusive) with first-episode psychosis. We will build on a Danish evidence-based intervention developed for young adults (OPUS) and adjust the concept to meet the specific needs of children and adolescents with early onset psychosis (OPUS YOUNG). The OPUS treatment is a coordinated and integrated manualized multimodal treatment building on three core elements: modified assertive community treatment with a low patient-case manager ratio; psychoeducational family intervention; and social skills training (SST). In OPUS YOUNG we will adjust the OPUS program to fit our younger age group by: 1) intensifying the support for caretakers and relatives including siblings, 2) instead of SST we are introducing social cognition and interaction treatment (SCIT), 3) providing individual cognitive behavioural case management (CBCM) to all participants and cognitive behavioural therapy (CBT) when needed, 4) addressing the specific challenges of psychopharmacologic treatment in adolescents by providing a treatment algorithm, 5) providing intensive supported transition of care (when patients approach transition to adult mental health services), 6) providing individualized school support, and 7) providing integrated prevention and treatment of substance misuse. Based on sample size estimation, we will include a minimum of 284 participants (maximum 304) and randomize them 1:1 to a two-year intervention of OPUS YOUNG versus TAU. We will conduct blinded assessment of treatment effects after 12 months and at treatment endpoint at 24 months. A further follow-up assessment will be performed to evaluate the sustainability of the intervention effects at six months after transition from OPUS YOUNG to TAU. Our primary outcome at treatment endpoint will be social function measured with Personal and Social Performance Scale (PSP). Secondary key outcomes measures are positive and negative symptoms, client satisfaction, and health related quality of life. Further outcomes are the broader psychopathology, cognitive functioning, social cognition, self-efficacy, experience of service, treatment alliance and adherence, the use of pharmacotherapy, school adherence, family burden, siblings' perceived stress, substance misuse, adverse treatment effects, and health economic measures.

ELIGIBILITY:
Inclusion Criteria:

1. Between 12 and 17 years of age (both inclusive) at trial inclusion.
2. First-episode psychosis within F2 spectrum (F20 schizophrenia, F21 Schizotypal disorder, F22 delusional disorder, F23 acute and transient psychotic disorders, F25 schizoaffective disorders, F28/29 other or un-specified non-organic psychosis) or depression with psychotic symptoms (F32.3, F33.3) or substance-induced psychosis (F1X.5) according to the International Statistical Classification of Diseases and Related Health Problems (ICD-10).
3. Maximum 12 months since first prescription of antipsychotic treatment on the indication psychosis.
4. Speak and understand Danish.
5. Written informed consent from parents or legal caretakers. Participants who reach age 18 years during the trial will be asked to give personal written informed consent to continue their study participation.

Exclusion Criteria:

1. A diagnosis of mental retardation of at least moderate severity defined as an intelligence quotient (IQ)of 49 or below (F71, F72, F73 according to the International Statistical Classification of Diseases and Related Health Problems (ICD-10).
2. Currently compulsory admission and/or treatment according to Danish legislation

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 284 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Personal and Social Performance Scale (PSP) | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Change in the global score of social function, measured with Personal and Social Performance Scale (PSP). PSP provides a global score on a scale from 1-100, with lower scores indicating lower social functioning. The global score is based on scores on four subdomains (1. Socially useful activities, 2. Personal and social relationships, 3. Self-care, and 4. Disturbing and aggressive behaviour), rated on a 6-point Likert scale (1=absent to 6=very severe). The scoring of PSP is based on all available information and concerns the patient's daily level of functioning in the family, in school, and during leisure time during the past month. Higher global values mean better social function. Researchers will interview the participants prior to the scoring of PSP using a semi structured interview guide suitable for children and adolescents, developed by the OPUS YOUNG research team.

SECONDARY OUTCOMES:
Severity of psychotic symptom dimension, SAPS | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Scale for Assessing Psychotic Symptoms in Schizophrenia (SAPS), used to assess the phenomenological presentation of psychotic symptoms in schizophrenia, is a rating scale to measure positive symptoms in schizophrenia. The SAPS- scale is split into 4 sub-scales (hallucinations, delusions, bizarre behavior and formal thought disorder) each of which are rated from 0 (absent) to 5 (severe) and for each domain is also given a global symptom severity score by the rater. The Psychotic symptom dimension is the sum of global scores, divided by the number of global scores (range 0-5). The psychotic dimension is composed of scores of hallucination and delusions. Higher score indicates worse level of symptoms.
Severity of Negative symptom dimension, SANS | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Scale for Assessing Negative Symptoms in Schizophrenia (SANS), used to assess the phenomenological presentation of negative symptoms in schizophrenia, is a rating scale to measure negative symptoms in schizophrenia. The SANS scale is divided into five sub-scales (affective flattening, alogia, avolition-apathy, anhedonia-asociality, attention), each of which are rated from 0 (absent) to 5 (severe) and for each domain is also given a global symptom severity score by the rater (global ratings). The Negative symptoms dimension is calculated as the sum of the global scores, divided by the number of global scores (range 0-5). The negative symptom dimension is composed of scores of anhedonia, avolition, affective flattening and alogia. Higher score indicates worse level of symptoms.
Severity of disorganized symptom dimension | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Severity of Disorganized symptom dimension is calculated as the sum of the global scores of formal thought disorder, bizarre and behaviors from Scale for Assessing Psychotic Symptoms in Schizophrenia (SAPS) and the score of inappropriate affects (item within the subscale for affective flattening) in Scale for Assessing Negative Symptoms in Schizophrenia (SANS) (range 0-5).Higher score indicates worse level of symptoms.
Client satisfaction questionnaire, CSQ | Present time at month 12 and at month 24.
  Patients satisfaction with the treatment is measured with the CSQ-scale. CSQ assess global client satisfaction, along with single dimension. The CSQ has eight question-items (quality of service, kind of service, met needs, recommend to a friend, amount of help, deal with problems, overall satisfaction, and come back). Patients respond to those question-items using a 4-point Likert scale. Their responses are scored from 1 to 4, and thus the possible total scores range from 8 to 32. Higher scores indicate greater satisfaction. Self-rapport
Quality of life, - Health Related Quality of Life Questionnaire for Children and Young People and their Parents, KIDSCREEN-10 | Last week at baseline (from enrollment), at month 12, at month 24 and at month 30
  The participants perception of their quality of life is assessed using the self-administered questionnaire KIDSCREEN-10. KIDSCREEN-10 contains 10 items: (1) Have you felt fit and well? (2) Have you felt full of energy? (3) Have you felt sad? (4) Have you felt lonely? (5) Have you had enough time for yourself? (6) Have you been able to do the things that you want to do in your free time? (7) Have your parent(s) treated you fairly? (8) Have you had fun with your friends? (9) Have you got on well at school? (10) Have you been able to pay attention? Participants respond to those question/items using a 5-point response scale. Answer categories item 1 and 9: not at all-slightly-moderately-very-extremely; all other items: never-seldom-quite often-very often-always. Responses are coded so that higher values indicate better QoL. A low score indicates a poor QOL, and a high score is indicative of a better QOL.

OTHER OUTCOMES:
Registration of multiaxial diagnostics, Schedule for affective disorders and schizophrenia for school-aged children (6-18 years) (K-SADS-PL), present and lifetime | Present and lifetime at baseline (from enrollment), at month 12 and at month 24
  Evaluation of clinical profile: by using K-SADS-PL scale for psychiatric diagnosis of patients.
Hallucinations, Experiences of thought disorder and Delusions, Schedules for Clinical Assessment in Neuropsychiatry (SCAN 2.1) | Present and lifetime at baseline (from enrollment), at month 12 and at month 24
  Hallucinations, Experiences of thought disorder and Delusions, measured with section 17 (Hallucinations), 18 (Experiences of thought disorder) and 19 (Delusions) in Schedules for Clinical Assessment in Neuropsychiatry (SCAN 2.1), using a rating scale (0 - 5), higher score indicating worse level of symptom.
Manic symptoms, (YMRS) | Last 2 days at baseline (from enrollment), at month 12, at month 24 and at month 30
  Young Maniac Rating Scale (YMRS), measure the severity of manic episodes. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. Total score rage is from 0 to 60 and the higher score represent a worse outcome.
Depressions, Hamilton-6, (HAM-6) | Last 3 days at baseline (from enrollment), at month 12, at month 24 and at month 30
  HAM-6 measures symptoms of depression for the last 3 days. Total score will be measured. Ranges from 0 to 22. Higher is worse.
Psychotic symptoms, Scale for Assessing Psychotic Symptoms in Schizophrenia (SAPS) | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Scale for Assessing Psychotic Symptoms in Schizophrenia (SAPS), clinician-administered questionnaire.The SAPS- scale is split into 4 sub-scales (hallucinations, delusions, bizarre behavior and formal thought disorder) each of which are rated from 0 (absent) to 5 (severe) and for each domain is also given a global symptom severity score by the rater (0 - 5). Higher score indicates worse level of symptoms.
Negative symptoms, Scale for Assessing Negative Symptoms in Schizophrenia (SANS) | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Scale for Assessing Negative Symptoms in Schizophrenia (SANS), clinician- administered questionnaire. Higher score indicates worse level of symptoms.The SANS scale is divided into five sub-scales (affective flattening, alogia, avolition-apathy, anhedonia-asociality, attention), each of which are rated from 0 (absent) to 5 (severe) and for each domain is also given a global symptom severity score by the rater (global ratings, range 0-5). Higher score indicates worse level of symptoms.
Global psychopathology, severity, The Clinical Impression Scale-Severity (CGI-S) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  The Clinical Impression Scale-Severity, (CGI-S), a clinician- administered scale for impression of global psychopathology, rated fra 1 (no sign of mental illness) to 7 (among the most extremely ill patients). Higher score indicates worse level of global Psychopathology.
Global psychopathology, Improvement, The Clinical Global Impression Scale - Improvement (CGI-I) | Last year at month 12, at month 24 and at month 30
  The Clinical Global Impression Scale - Improvement, (CGI-I), a clinician-administered scale for impression of global improvement of the patients mental health rated from 1(very much improved) to 7 (very much worse). Higher score indicates worse level mental health since the year before.
Suicidal behavior | Present and lifetime at baseline (from enrollment), at month 12, at month 24 and at month 30
  Self-reported suicidal ideation questionnaire, the patients answer yes or no to question of suicidal behavior ( whether they have ever had suicidal thoughts, and if so, how frequently and whether they acted on and what they did). Positive answer (Yes) means worse outcome.
Changes in global cognitive functioning, Brief Assessment of Cognition in Schizophrenia (BACS) | Present time at baseline (from enrollment) and at month 24
  The Brief Assessment of Cognition in Schizophrenia (BACS) includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. Z-scores are calculated from composite scores. Higher z-scores are indicative of better cognitive performance, lower z-scores are indicative of lower cognitive performance. Range of z-scores anticipated to be between -3 and 3.
Changes in social cognition, Hinting Task | Present time (from enrollment) and at month 24
  Hinting Task measures Theory of Mind
Changes in social cognition, EIMT | Present time (from enrollment) and at month 24
  Emotional Intensity Morphing Task (EIMT) measures facial emotional recognition
General self-efficacy (GSE) (patients) | Present time (from enrollment), at month 12, at month 24 and at month 30
  Measures general belief in one's own capabilities. Self-report. Total score is measured. Ranges from 10 to 40. Higher scores indicate better self-efficacy
Treatment alliance Working Alliance Inventory scale (WAI) | Last month at month 12, at month 24 and at month 30
  Measured the experience of alliance between the client and the therapist(s). Self-report. Total score is measured. Ranges from 12 to 60. Higher scores indicate better alliance.
Negative effects of psychological treatment questionnaire (NEQ) | Last 2 years at month 24
  Self-reported questionnaire of participants impressions of negative effects of the treatment they received. The NEQ answers 16 questions about their impressions of negative effects of the treatment, from 1 (not at all) to 5 (very much). Higher score means worse.
School adherence | Last 3 month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Days in school/education/employment, self-report
Quality-adjusted life year, European Quality of Life (EuroQol) 5-Dimension 5-Level (EQ 5D - 5L) Questionnaire General Health Status Score | Present time at baseline (from enrollment), at month 12, at month 24 and at month 30
  Self-reported questionnaire, EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The responses to the 5 dimensions are used to compute a single utility score ranging from zero (worst health state) to 1 (better health state) representing the general health status of the individual.
Children health, The Child Health Utility (CHU9D) | Present time at baseline (from enrollment), at month 12, at month 24 and at month 30
  Self-reported questionnaire about children's health consists of 9 items, each with 5 response categories (scored 1-5) that assess the child/adolescent functioning "today" across domains of worry, sadness, pain, tiredness, annoyance, school, sleep, daily routine and activities. The instrument is available in both self-report (completed by the child). Higher scores mean a worse outcome.
Substance abuse, Timeline Follow Back, Trivsel og effekt monitorering (TEM) | Last 4 weeks at baseline (from enrollment), at month 12, at month 24 and at month 30
  Measured using the Timeline Follow Back interview TEM, in which you systematically go through every day for the last 4 weeks recording any alcohol and drug (legal and illegal) consumption.
  Less consumed alcohol and substance will be considered better
Medication side-effects, (Danish scale for medication side-effects) Bivirkningsskala Skala Til Registering af Uønskede Virkninger af Psykofarmaka, UKU. | Last 3 days at baseline (from enrollment), at month 12, at month 24 and at month 30
  Registration and assessment of medication side-effects the last 3 days. Possible score: 0 (not present) to 3 (present to a severe degree). Higher scores mean worse outcome.
Self-reported use of antipsychotic medication | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  The use of antipsychotics and any other medication (drug, daily dosage, duration) will be carefully recorded in both the experimental group and the treatment as usual (TAU) group. Information on medication use will be obtained through the participant's medical journal and by self-reported information at the assessment interview.
Executive Function, Behavior Rating Inventory of Executive, 2. edition (BRIEF-2), parent reported questionnaire. | Last six month at baseline (from enrollment), at month 12, at month 24 and at month 30
  A questionnaire for parents to assess executive functions, the BRIEF-2, Parent Form is used for children and young people aged 5-18 years and it includes 63 statements about the child's behavior in everyday life. The statements of BRIEF-2 have 3 (force-choice) possible answers: never (score of 1), sometimes (score of 2), often (score of 3);. The BRIEF-2 includes clinical subscales that measure different aspects of executive functions such as Inhibit, Self-Monitoring, Flexibility, Emotional Control, Initiation, Working Memory, Planning / Organizing, Task Monitoring, and Organizing Materials. Based on these subscales, the BRIEF-2 generates 3 indices (Behavior Regulation, Emotion Regulation, and Cognitive Regulation) as a Global Executive Functioning measure. The Global Executive Functioning raw scores range from a minimum 60 to maximum of 180. Higher scores mean worse executive problems.
Parental stress (PSS) parent reported questionnaire. | Present and lifetime at baseline (from enrollment), at month 12, at month 24 and at month 30
  The parental stress scale is a parent-reported questionnaire (range 18 -90), a higher score indicates more parental stress
Family function (FAD) | Present time at baseline (from enrollment), at month 24 and at month 30
  60-item self-report measure of family functioning answered on a four-point Likert scale ranging from 'strongly agree' to 'strongly disagree'.
General self-efficacy (GSE) parent-reported questionnaire. | Present time (from enrollment), at month 12, at month 24 and at month 30
  Measures general belief in one's own capabilities. Total score is measured. Ranges from 10 to 40. Higher scores indicate better self-efficacy
The Client satisfaction questionnaire (CSQ). Parent-reported questionnaire. | Present time at month 12 and at month 24
  Measures satisfaction with treatment. Total score is measured, ranging from 8 to 32. Higher scores indicate higher satisfaction. Self-report
Negative effects of psychological treatment (NEQ). Parent-reported questionnaire. | Last 2 years at month 24
  Self-reported questionnaire of parents impressions of negative effects of the treatment. The NEQ has 16 questions about their impressions of negative effects of the treatment, from 1 (not at all) to 5 (very much). Higher score means worse.
Use of psychopharmacological treatment | From the participant enters the study to month 30
  Individual-level data retrieved from The National Patient Register, containing information about contacts with the health care system during the trial period. Data is routinely collected in the Danish health care system independent of this present study. Contacts with the health care system will be assessed and compared as incidence rates of acute/non acute, in-patient/outpatient and psychiatric/somatic contacts.
Register-based information (others) | At 30 months (6 months follow-up after end-of-trial)
  Data on the patients will be extracted from the following registers from Statistics Denmark: The Danish Population Register, the Danish Psychiatric Central Register, the Danish Education Register, the Danish Register of Special Education, the Danish Institution Register, the Danish Register of School Grades, the Danish Patient Register, the Danish Prescription Register, and the Danish Migration Register. We will assess socio-demographic information including school attendance, school grades and exams, labour market affiliation, civil status, cohabitation status, data on complications to the pregnancy and birth of the participant, education, living in an institution (and type of institution), use of any health care and social services and, in the unlikely event: cause of death.
Electrocardiogram (ECG), standard leads | Present and at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record.
Personal and Social Performance Scale (PSP), subdomains | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Subdomains of the PSP. PSP is a validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point Likert scale (1=absent to 6=very severe), . The scoring of PSP is based on all available information and concerns the patient's daily level of functioning in the family, in school, and during leisure time during the past month. Researchers will interview the participants prior to the scoring of PSP using a semi structured interview guide suitable for children and adolescents, developed by the OPUS YOUNG research team. Higher score indicating worse function
Use of health care services | Last month at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from Danish National Patient Register containing information about contacts with the health care system during the follow-up period. Data is collected routinely in the Danish health care system, independent of this present study. Contacts with the health care system will be assessed and compared as incidence rates of acute/non-acute, in-patient/out-patient and psychiatric/somatic contacts.
Triglycerides | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record. Measurement of lipids (in serum), triglycerides (mmol/l)
Total cholesterol | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record. Measurement of lipids (in serum), total cholesterol,(mmol/l)
Low density lipoprotein (LDL) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record. Measurement (mmol/l) of lipids (in serum), low density lipoprotein ( LDL), (mmol/l)
Very-low-density lipoprotein (VLDL) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record. Measurement of lipids (in serum), very-low-density lipoprotein (VLDL), (mmol/l)
High density lipoprotein, (HDL) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record. Measurement of lipids (in serum), high density lipoprotein (HDL), (mmol/l)
Glucose values | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record. Fasting glucose values, blood test, (mmol/L)
Determination of prolactin | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record. Determination of prolactin, blood test, (nmol/l)
Haemoglobin | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, red blood cell status, haemoglobin, blood test (mmol/l)
Leukocyte cell count (and differential count) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patient's' medical record, white blood cell status, leukocyte cell count (and differential count), (x 10/l) blood test.
Thrombocyte cell count | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, thrombocyte cell count(x 10/l) blood test.
Sodium (Na) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, electrolytes, sodium (Na), blood test (mmol/l)
Potassium (Ka) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, electrolytes, potassium (Ka), blood test (mmol/l)
Creatinine | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, electrolytes, creatinine, blood test (micromol/l)
Aspartate transaminase, (ASAT) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, Liver test: aspartate transaminase, (ASAT), blood test (U/l)
Alkaline phosphatases; | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, Liver test: alkaline phosphatases, blood test (U/l)
Thyroid-stimulating hormone (TSH) | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, metabolism: thyroid - stimulating hormone (TSH), blood test (mU/l)
Vitamin D | Present at baseline (from enrollment), at month 12, at month 24 and at month 30
  Individual-level data retrieved from the patients' medical record, vitamin D, (nmol/l), blood test

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Pagsberg, PhD, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Mental Health Services in the Capital Region, Denmark, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No
The investigators will share the depersonalized data at www.clinical Trials.gov

REFERENCES:
- [Derived] Madsen MS, Melau M, Andersen NK, Nielsen CF, Larsen N, Andersen TL, Nordentoft M, Jepsen JRM, Thorup AAE, Jeppesen P, Fagerlund B, Rimvall MK, McGorry P, Singh S, Vernal DL, Hastrup LH, Olsen LR, Rydkjaer J, Correll CU, Christensen R, Pagsberg AK. Early intervention versus treatment as usual for adolescents with first-episode psychosis: Protocol for the randomized OPUS YOUNG trial. Contemp Clin Trials. 2026 Feb 5:108253. doi: 10.1016/j.cct.2026.108253. Online ahead of print. PMID 41654084

DOCUMENTS (1):
  • Study Protocol (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT04916626/Prot_000.pdf